CLINICAL TRIAL: NCT02959788
Title: Heart Rate Variability as a Predictor of Ischemic Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Mohr, Nicholas M, Associate Professor, University of Iowa
Other Study IDs: 201512751
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Heart rate variability
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain patients: All patients who present to the ED with chest pain.
  Interventions: Other: Heart rate variability

INTERVENTIONS:
Other: Heart rate variability — All patients have a 10-minute recording analyzed for indices of heart rate variability.

SUMMARY:
Identification of patients who are at highest risk for heart attack is an important task for emergency medicine physicians. Currently, physicians use a variety of different scoring systems to stratify their risk for having a heart attack. Heart rate variability (HRV) is a measure derived from noninvasive cardiac monitoring. This data is collected from a simple, non-invasive chest strap during a 10-minute recording session. The purpose of this proposal is to collect heart rate variability data on patients admitted to the emergency department with chest pain. The intent is to measure the association between heart rate variability and the various risk stratification scoring systems for chest pain.

DETAILED DESCRIPTION:
Identification of patients who are at highest risk for heart attack is an important task for emergency medicine physicians. Currently, physicians use a variety of different scoring systems to stratify their risk for having a heart attack. Heart rate variability (HRV) is a measure derived from noninvasive cardiac monitoring. This data is collected from a simple, non-invasive chest strap during a 10-minute recording session. The purpose of this proposal is to collect heart rate variability data on patients admitted to the emergency department with chest pain. The intent is to measure the association between heart rate variability and the various risk stratification scoring systems for chest pain.

The investigators propose to enroll patients admitted to the emergency department with chest pain. In addition to HRV data, clinical risk factors will be obtained, using validated clinical risk scoring systems. The team will follow patient's clinical course in order to include information about the determined cause of chest pain. The goal is to understand how HRV can augment common risk stratification scoring systems for patient presenting to the ED with chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain in ED

Exclusion Criteria:

* STEMI
* Prisoners
* Pregnant women
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults who present to the emergency department with chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 30 days

SECONDARY OUTCOMES:
HEART score | 1 day
Coronary heart disease risk factors | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Mohr, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No